CLINICAL TRIAL: NCT06075693
Title: Cerebrospinal Fluid Biomarkers of Myotonic Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thurman Wheeler, M.D, Physician Scientist, Massachusetts General Hospital
Other Study IDs: 2021P002482; U01FD008128 (FDA)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Myotonic Dystrophy Type 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Longitudinal: We will ask eligible volunteers to provide a CSF sample by a lumbar puncture procedure, a urine sample, undergo a cognitive assessment, and to undergo an MRI scan once per year for two years.
- Single: We will ask eligible volunteers to provide a CSF sample by a lumbar puncture procedure, a urine sample, undergo a cognitive assessment, and to undergo an MRI scan once.

SUMMARY:
Myotonic dystrophy is associated with central sleep apnea, excessive daytime sleepiness, diminished working memory, impaired visuospatial skills, and deficits in problem-solving skills.

Cerebrospinal fluid (CSF) is a clear, colorless fluid that surrounds and protects the brain.

Changes in the composition of CSF can serve as early indicators of changes in brain activity and function. The purpose of this research is to learn about myotonic dystrophy by examining cerebrospinal fluid and brain activity in participants. The tests will be low risk and are well tolerated. The information that we gather from this study may help us evaluate, prevent, diagnose, treat, and improve our understanding of myotonic dystrophy. Funding Source- FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Subjects with DM1 based on genetic testing and/or clinical criteria (some subjects who have positive genetic testing may be asymptomatic, while other subjects who show characteristic clinical features may have declined to have genetic testing done).
* Unaffected subjects are unknown to have myotonic dystropphy or any other muscular dystrophy by history and may have had no genetic testing.
* Clinical indicators of current status, as measured within 30 days of study start: Able to provide informed consent or assent for participation in the study.
* Demographic characteristics (e.g., biologic sex, age): Males and females age 18 years and older.

Exclusion Criteria:

* Medical history of any of the following. State of immunosuppression; pre-existing liver or kidney disease; documented HIV positive; documented hepatitis B and/or C positive.
* Medications and other drugs. Use of anticoagulants within 60 days prior to lumbar puncture and/or blood draw. Use of anti-platelet drugs within 7 days prior to blood draw.
* Contraindications to MRI. The presence of any metal within the body, which would include any medical device containing metal, such as a pacemaker, defibrillator, some heart valves or stents, artificial joint, aneurysm clip, or inner ear device, a history of working with sheet metal, or an injury with metal shrapnel; pregnancy, due to effects of MRI on unborn children.
* Contraindications to Lumbar Puncture. Evidence of increased intracranial pressure or active infection on exam; platelets less than 50,000.
* Other. Inability or unwillingness of the subject to give written informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Individuals with myotonic dystrophy type 1 (DM1), ages 18 and older.
  2. Individuals without myotonic dystrophy (unaffected), ages 18 and older.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Extracellular RNA splice variants in biofluids | 5 years
  The extracellular RNA biomarkers in the muscular dystrophy groups will be evaluated and compared with the extracellular RNA content in control groups. Statistical analysis will be used to evaluate the sensitivity and specificity of these markers as measurements of disease activity and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Thurman M Wheeler, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No